CLINICAL TRIAL: NCT00003451
Title: Phase I Trial of Interleukin-12 Followed by Interferon-Alpha
Brief Title: Interleukin-12 Followed by Interferon Alfa in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01397; OSU-T98-0020; NCI-T98-0020; CDR0000066482 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage III multiple myeloma; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Interferon-alpha; Interleukin-12 Subunit p35

ARMS (1):
- Arm I (Experimental): Cohorts of 3 patients receive interleukin-12 IV push on day 1, followed by escalating doses of interferon alfa by subcutaneous injection at 24, 48, 72, 96 and 120 hours. Courses repeat every 2 weeks for 6 months (12 courses total) in the absence of unacceptable toxicity and disease progression. Patients achieving partial response or stable disease at the completion of 6 months of therapy may receive additional courses of therapy for up to 24 months. Dose escalation of interferon alfa continues in subsequent cohorts in the absence of dose limiting toxicity (DLT). If 1 of 3 patients experiences DLT at a dose level, then 3 additional patients are entered at that dose level. If 2 of 6 patients experience DLT, then dose escalation stops. The maximum tolerated dose is defined as 1 level below that dose at which 2 or more of 6 patients experience DLT. Patients are followed every 3 months for 1 year and then every 6 months thereafter.
  Interventions: Biological: recombinant interferon alfa; Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: recombinant interleukin-12

SUMMARY:
Phase I trial to study the effectiveness of combining interleukin-12 and interferon alfa in treating patients who have residual, recurrent, or metastatic malignant melanoma or other advanced cancer that has not responded to standard therapy. Interleukin-12 may stimulate a person's white blood cells to kill cancer cells. Interferon alfa may interfere with the growth of the cancer cells. Combining interleukin-12 with interferon alfa may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of interferon alfa when preceded by a single dose of interleukin-12 in patients with recurrent or metastatic melanoma or other advanced malignancies.

OUTLINE: This is a dose-escalation study.

Cohorts of 3 patients receive interleukin-12 IV push on day 1, followed by escalating doses of interferon alfa by subcutaneous injection at 24, 48, 72, 96 and 120 hours. Courses repeat every 2 weeks for 6 months (12 courses total) in the absence of unacceptable toxicity and disease progression. Patients achieving partial response or stable disease at the completion of 6 months of therapy may receive additional courses of therapy for up to 24 months. Dose escalation of interferon alfa continues in subsequent cohorts in the absence of dose limiting toxicity (DLT). If 1 of 3 patients experiences DLT at a dose level, then 3 additional patients are entered at that dose level. If 2 of 6 patients experience DLT, then dose escalation stops. The maximum tolerated dose is defined as 1 level below that dose at which 2 or more of 6 patients experience DLT. Patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed residual, recurrent, or metastatic malignant melanoma or other advanced malignancies
* Must have failed standard curative and/or palliative therapies
* No brain or central nervous system metastases

PATIENT CHARACTERISTICS:

* Age: 13 and over
* Performance status: Karnofsky 70-100%
* Life expectancy: At least 12 weeks
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (may be posttransfusion or may receive erythropoietin)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min
* Calcium no greater than 11 mg/dL (may receive agents to decrease calcium)
* No significant cardiovascular disease
* No cardiac arrhythmia requiring drug or device intervention
* No history of significant peripheral neuropathy
* No significant central nervous system disease
* HIV negative Hepatitis B surface antigen negative
* No concurrent serious infection requiring intravenous antibiotic therapy
* No clinically significant autoimmune disease (i.e., rheumatoid arthritis)
* No clinically significant gastrointestinal bleeding or uncontrolled peptic ulcer disease
* No history of inflammatory bowel disease
* No other major illness that substantially increases the risk associated with participation in this study
* Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior biologic therapy
* At least 4 weeks since prior chemotherapy
* No concurrent systemic corticosteroids
* At least 2 weeks since prior local radiotherapy
* At least 2 weeks since surgery Other: At least 4 weeks since prior investigational drug

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-08; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E. Carson, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States